CLINICAL TRIAL: NCT06968715
Title: The Effects of 12-week Hydrogen-rich Water Consumption on Body Composition and Metabolic Biomarkers in Adults With Metabolic Syndrome and Varying Breath Hydrogen Levels
Brief Title: Hydrogen-Rich Water and Metabolic Health in Adults: A 12-Week Randomized Trial
Acronym: HYDRO-RESPOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 51-02-01
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental 1: low-breath hydrogen (Experimental): One liter of hydrogen-rich water per day
  Interventions: Dietary Supplement: Experimental 1: low-breath hydrogen
- Experimental 2: high-breath hydrogen (Experimental): One liter of hydrogen-rich water per day
  Interventions: Dietary Supplement: Experimental 2: high-breath hydrogen
- Experimental 3: low-breath hydrogen (Placebo Comparator): One liter of control water per day
  Interventions: Dietary Supplement: Experimental 3: low-breath hydrogen
- Experimental 4: high-breath hydrogen (Placebo Comparator): One liter of control water per day
  Interventions: Dietary Supplement: Experimental 4: high-breath hydrogen

INTERVENTIONS:
Dietary Supplement: Experimental 1: low-breath hydrogen — Hydrogen-rich water (1.0 L/day)
  Arms: Experimental 1: low-breath hydrogen
Dietary Supplement: Experimental 2: high-breath hydrogen — Hydrogen-rich water (1.0 L/day)
  Arms: Experimental 2: high-breath hydrogen
Dietary Supplement: Experimental 3: low-breath hydrogen — Placebo water (1.0 L/day)
  Arms: Experimental 3: low-breath hydrogen
Dietary Supplement: Experimental 4: high-breath hydrogen — Placebo water (1.0 L/day)
  Arms: Experimental 4: high-breath hydrogen

SUMMARY:
The HYDRO-RESPOND trial is a 12-week randomized controlled study investigating the effects of daily hydrogen-rich water (HRW) consumption on body composition and metabolic biomarkers in adults diagnosed with metabolic syndrome. The study also explores whether individual differences in baseline breath hydrogen levels influence response to HRW. Participants are randomly assigned to receive either HRW or a placebo, with outcomes including changes in body fat, waist circumference, glucose metabolism, lipid profiles, and inflammatory markers. The trial aims to determine the therapeutic potential of HRW and identify predictors of individual responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-65 years
* Metabolic syndrome (NHS) (at least 3 of the 5 following criteria):

  * Waist circumference of ≥ 102 cm in men and ≥ 88 cm in women
  * Hypertriglyceridemia (≥ 1.695 mmol/L)
  * Low HDL-C (< 1.04 mmol/dL in men and < 1.30 mmol/dL in women)
  * High blood pressure (> 130/85 mmHg)
  * High fasting glucose (> 6.1 mmol/L)
* Not physically active
* Informed consent signed

Exclusion Criteria:

* Major chronic disease and acute injuries
* History of dietary supplement use during the past 4 weeks
* History of metabolism-modulating pharmaceuticals use during the past 4 weeks
* No consent to randomization
* Participation in other studies

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Waist circumference | Change from baseline waist circumference at 12 weeks
  Waist circumference, measured at the midpoint between the lower rib and iliac crest, serves as an indicator of abdominal adiposity and a key outcome reflecting metabolic risk.

SECONDARY OUTCOMES:
Body fat | Change from baseline body fat at 12 weeks
  Body fat measured with bioimpedance analysis
Lipoprotein (a) | Change from baseline lipoprotein (a) at 12 weeks
  Serum levels of lipoprotein (a)
Total antioxidant capacity | Change from baseline total antioxidant capacity at 12 weeks
  Serum levels of total antioxidant capacity

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Bioenergetics Lab at Faculty of Sport and PE, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in metabolic syndrome. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Only qualified researchers with academic interest in metabolic syndrome or molecular hydrogen research